CLINICAL TRIAL: NCT06760975
Title: Comparative Effects of Vestibular Habituation and Ocular Reflex Exercises on Gait Stability, Dizziness Severity, and Fear of Fall in Elderly Population With Vertigo
Brief Title: Effects of Vestibular Habituation and Ocular Reflex Exercises on Vertigo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0255
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Vertigo
Keywords: vertigo; Habituation; Ocular reflex; Fear of fall; Gait stability
MeSH Terms: conditions — Vertigo; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as Assessor of the study would be kept blind of the treatment groups to which patient will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A Vestibular Habituation Exercises (Experimental): Group A will receive 24 sessions of vestibular habituation exercises, delivered 4 times weekly for six weeks, each session lasting 30 minutes. Effects will be measured at baseline, in the 3rd week, post-intervention, after six weeks, and at a 9th-week follow-up.
  Interventions: Other: Vestibular Habituation Exercises
- GROUP B Ocular Reflex exercises (Experimental): Group B will receive ocular reflex exercises. A total of 24 sessions (4x/week for 6 weeks) will be conducted , lasting 50-60 minutes each. The effects will be measured at baseline, in the 3rd week, post intervention, after six weeks, and at a 9th-week follow-up.
  Interventions: Other: Ocular Reflex Excercises

INTERVENTIONS:
Other: Vestibular Habituation Exercises — The vestibular habituation exercise group follows a structured progression over six weeks. in week 1 participants perform large amplitude, rapid cervical rotations seated, completing 3 sets of five cycles each. By week 2, the exercises increase in complexity , incorporates standing pivots or seated trunk flexion extension. in week 3 the cervical rotations are continued with seated or standing posture. week 4 introduces a busy visual background during the exercise to challenge visual-vestibular integration. In week 5 the exercises are performed standing with the addition complex visual target against a busy background. finally week 6 includes most advance movement including standing pivots 180 degrees and brand-daroff exercises with further visual challenges of near and far targets in busy background. Each exercise session last for 2 minutes and is aimed at progressively enhancing vestibular processing and adaptability.
  Arms: GROUP A Vestibular Habituation Exercises
Other: Ocular Reflex Excercises — The Ocular reflex exercises focuses on enhancing visual tracking and reflexes through targeted viewing exercises. In week 1, participants perform horizontal and vertical X1 viewing exercises with a near target, holding each position for 1 minute while seated. In week 2 the duration of the X1 exercises is extended to 2 minutes with the near target still in seated position. Week 3 shift to a far target for the X1 exercises and the participants performs them while standing increasing the challenge. By week 4 the exercise incorporate both near and far target in front of a busy background. extending the duration to 2 minutes while standing. In week 5 horizontal and vertical X2 viewing exercises are added with a plain background, while still using near and far targets in front of a busy background . finally week 6 continues the X1 and X2 exercises with near and far targets in a busy background, performed for 2 minutes while standing. This aims to improve visual tracking.
  Arms: GROUP B Ocular Reflex exercises

SUMMARY:
The aim of this study is to determine the comparative effects of vestibular Habituation and ocular reflex exercises on Gait stability, Dizziness severity, and fear of fall in elderly population with vertigo

DETAILED DESCRIPTION:
vestibular habituation exercises focus on helping individual adapt to and reduce symptoms related to vestibular disorder such as improving balance , reducing dizziness and enhance overall functional abilities. ocular reflex exercises focus on improving eye movement control and coordination such as improving visual tracking , stability and Focus. This randomized clinical trial will be conducted at services hospital and Jinnah hospital for a duration of 10 months. The sample size will consist of 50 participants. 25 participants will be assigned to vestibular habituation exercise group and 25 to ocular reflex exercises group. Data will be collected using these assessment tools, including the dynamic gait index for gait stability, the fall efficacy scale for fear of fall, and dizziness handicap inventory for dizziness severity. Pre-intervention assessments will be conducted for all two groups. The effects of the interventions will be measured at baseline ,in the 3rd week ,post intervention, after 6 weeks, and at a 9th week follow up. Data analysis will be performed by using SPSS 26 software

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients
2. Age 65-75
3. patient with vestibular disorder for at least 6 months
4. patient with unspecific dizziness sensation for at least 3 months
5. Dizziness handicap inventory score > 16 -

Exclusion Criteria:

1. patient with central nervous system diseases, like stroke, multiple sclerosis, Parkinson's disease.
2. orthopedic problems that precluded performance of the exercises
3. systemic diseases with no medication control
4. if patient were legally blind or had dementia
5. patient with no history of epilepsy and other neurological diseases -

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Dynamic gait index | 6 weeks
  The DGI is used for gait assessment and has 8 items. The scoring of DGI is based on 4 point scale ranging from 0-3 while 0 indicates severe impairment and 3 indicates normal ability. DGI proves to be reliable and valid for older people. Total score for best performance is 24 and low score on DGI indicates greater impairment in functional mobility.
FES-I Fall efficacy scale international | 6 weeks
  FES-I scale is used to access fear of fall and is consist of 16 items questionnaire allows participants to rate their fear of falling during specific activities at the rate of four different intensities ranging from "not at all concerned to vary concerned". Higher scores indicates a more significant fear of falling. score range from 16-19 show low concern of falling. Score ranges from 20-27 shows moderate concern and score ranges from 28-64 show high concern of fall to daily Activities.
Dizziness Handicap inventory | 6 weeks
  The DHI is used to access dizziness and is consist of 25 items. Each item is answered with No (0) points sometimes (2) points or Yes (4) points. Scoring of DHI ranges from 0 to 100. further divided into physical (28) points , functional (36) points and emotional (36) points. The higher the scores result in perceived handicap. Moreover (DHI) proved to be a reliable instument

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, MS-NMPT, Study Chair — Riphah International University
Locations (2):
- Pakistan (2):
  - Rasheed Hospital Lahore, Lahore, Punjab Province
  - Services Hospital Lahore, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayat A, Pourbakht A, Saki N, Zainun Z, Nikakhlagh S, Mirmomeni G. Vestibular rehabilitation outcomes in the elderly with chronic vestibular dysfunction. Iran Red Crescent Med J. 2012 Nov;14(11):705-8. doi: 10.5812/ircmj.3507. Epub 2012 Nov 15. PMID 23396380
- [Background] Balatsouras DG, Koukoutsis G, Fassolis A, Moukos A, Apris A. Benign paroxysmal positional vertigo in the elderly: current insights. Clin Interv Aging. 2018 Nov 5;13:2251-2266. doi: 10.2147/CIA.S144134. eCollection 2018. PMID 30464434
- [Background] Cohen HS, Kimball KT. Increased independence and decreased vertigo after vestibular rehabilitation. Otolaryngol Head Neck Surg. 2003 Jan;128(1):60-70. doi: 10.1067/mhn.2003.23. PMID 12574761
- [Background] Hall CD, Heusel-Gillig L, Tusa RJ, Herdman SJ. Efficacy of gaze stability exercises in older adults with dizziness. J Neurol Phys Ther. 2010 Jun;34(2):64-9. doi: 10.1097/NPT.0b013e3181dde6d8. PMID 20588090
- [Background] Norre ME, Beckers A. Vestibular habituation training: exercise treatment for vertigo based upon the habituation effect. Otolaryngol Head Neck Surg. 1989 Jul;101(1):14-9. doi: 10.1177/019459988910100104. PMID 2502758
- [Background] Strupp M, Brandt T. Diagnosis and treatment of vertigo and dizziness. Dtsch Arztebl Int. 2008 Mar;105(10):173-80. doi: 10.3238/arztebl.2008.0173. Epub 2008 Mar 7. PMID 19629221